CLINICAL TRIAL: NCT00043225
Title: Clinical Course in Cystic Fibrosis: The Effects of Pseudomonas Aeruginosa and Potential Modifier Genes
Brief Title: The Role of Bacteria and Genetic Variations in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010198; 01-H-0198
Record Dates: First submitted 2006-07-13; First posted 2002-08-07 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Psuedomas Infection; Cystic Fibrosis
Keywords: Type III Secretion Pathways; Exotoxin A Polymorphisms; Cystic Fibrosis and Pseudomonas Aeruginosa; Adenosine Deaminase Deficiency; Severe Combined Immune Deficiency; SCID; ADA-SCID; Immune Deficiency
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections; Severe combined immunodeficiency due to adenosine deaminase deficiency; Severe Combined Immunodeficiency; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cystic Fibrosis: Cystic Fibrosis patients

SUMMARY:
This study will examine 1) the role of hereditary factors in cystic fibrosis; i.e., the relationship of the disease to specific gene variations, and 2) the role of bacterial products involved in lung infections substances produced by bacteria may worsen the disease.

Patients with cystic fibrosis who are being followed by the Medical College of Wisconsin or the University of Wisconsin-Madison are eligible for this study. Participants will have blood tests, pulmonary function tests, a sputum culture, and buccal swabbing (cotton swabbing of the inside of the cheek to collect cells for DNA study). In addition, their medical records will be reviewed for a history of lung infections and the results of various tests, including pulmonary function studies, chest X-rays and bacterial cultures. Blood samples collected previously at the Medical College of Wisconsin or the University of Wisconsin-Madison will also be analyzed for antibodies to bacteria.

Although this is a one-time study, participants may be asked to return for repeated tests.

...

DETAILED DESCRIPTION:
Individuals with cystic fibrosis (CF) are susceptible to chronic bacterial colonization by Pseudomonas aeruginosa, which results in deterioration of lung function and, eventually, death. In this study, we hope to improve our understanding of the innate immune response to infection by strains of P. aeruginosa that express type III cytotoxins and to delineate better the role of modifier genes in disease progression.

We will examine relationships between the patient's clinical course, the presence of antibodies to P. aeruginosa, and single nucleotide polymorphisms in suspected CF modifier genes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with cystic fibrosis who have a defined mutation in CFTR (e.g., any of the known variants of the CFTR gene, such as the delta F508 allele) born in the state of Wisconsin since 1985 or otherwise followed by the cystic fibrosis centers at the Medical College of Wisconsin or University of Wisconsin-Madison.

Patients will have been tested or will be tested for the CFTR gene under another protocol (96-H-0100).

Patients may be colonized with P. aeruginosa or other organisms (e.g., Burkholderia cepacia).

The age range of NIH participants in this study is from 9 to 80 years old.

EXCLUSION CRITERIA:

There are no exclusion criteria.

Ages: 9 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with cystic fibrosis (CF) are susceptible to chronic bacterial colonization by @@@Pseudomonas aeruginosa, which results in deterioration of lung function and, eventually, death. In this study, we hope to improve our understanding of the innate immune response to infection by strains of P. aeruginosa that express type III cytotoxins and to delineate better the role of modifier genes in disease progression.@@@
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2001-06-20 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
There is a relationship between the virulence characteristics of P.aeruginosa involved inpersistent infection of the lung and the genetic profile of CF patients. | End of study
  There is a relationship between the virulence characteristics of P.aeruginosa involved in persistent infection of the lung and the genetic profile of CF patients.

SECONDARY OUTCOMES:
Antibodies to the components of the type III secretion pathway can be used as an accurate measure of acute infection and colonization of the CF lung by virulent strains of P. aeruginosa. There is a relationship between modifier genotypes and sur... | End of Study
  Antibodies to the components of the type III secretion pathway can be used as an accurate measure of acute infection and colonization of the CF lung by virulent strains of P. aeruginosa. There is a relationship between modifier genotypes and survival or other measurable CF disease outcomes. 4. The bactericidal activity of sera from CF patients will neutralize components of the Type III pathway

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (4):
- United States (4):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Riordan JR, Rommens JM, Kerem B, Alon N, Rozmahel R, Grzelczak Z, Zielenski J, Lok S, Plavsic N, Chou JL, et al. Identification of the cystic fibrosis gene: cloning and characterization of complementary DNA. Science. 1989 Sep 8;245(4922):1066-73. doi: 10.1126/science.2475911.
- [Background] Rommens JM, Iannuzzi MC, Kerem B, Drumm ML, Melmer G, Dean M, Rozmahel R, Cole JL, Kennedy D, Hidaka N, et al. Identification of the cystic fibrosis gene: chromosome walking and jumping. Science. 1989 Sep 8;245(4922):1059-65. doi: 10.1126/science.2772657.
- [Background] Frizzell RA. Functions of the cystic fibrosis transmembrane conductance regulator protein. Am J Respir Crit Care Med. 1995 Mar;151(3 Pt 2):S54-8. doi: 10.1164/ajrccm/151.3_Pt_2.S54. PMID 7533606
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-H-0198.html